CLINICAL TRIAL: NCT05303194
Title: Patient Priorities Care for Hispanics With Dementia
Acronym: PPC-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0107
Record Dates: First submitted 2022-03-08; First posted 2022-03-31 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Multiple Chronic Conditions; Dementia
Keywords: multiple chronic conditions; dementia; Hispanic
MeSH Terms: conditions — Multiple Chronic Conditions; Dementia

STUDY DESIGN:
Intervention Model Description: The study has two phases: 1) an initial adaptation phase; and 2) a feasibility testing phase. For the adaptation phase 5 Hispanics with multiple chronic condition and without dementia will be invited to participate. These participants will need to consent to be part of the study. For the second phase, the investigators will determine if participants with dementia have capacity by asking their primary care providers or by administering the telephone version of the Montreal Cognitive Assessment. If a score of less than 12 is obtained, the caregiver will be asked to consent for both participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Priorities Care (PPC) Adaptation (Other): 5 Hispanic patients with multiple chronic conditions (MCC) and no dementia. In order to adapt PPC for Hispanics with MCC, five Hispanics with MCC will go through the 2 parts of the PPC approach: 1) Priority setting; and 2) Care alignment.
  Interventions: Behavioral: Patient Priorities Care (PPC) Approach
- PPC Feasibility Testing (Other): 20 Hispanic patients with multiple chronic conditions (MCC), including dementia. In order to adapt PPC for Hispanics with MCC and dementia, twenty Hispanics with MCC and dementia will go through the 2 parts of the PPC approach: 1) Priority setting; and 2) Care alignment.
  Interventions: Behavioral: Adapted PPC

INTERVENTIONS:
Behavioral: Patient Priorities Care (PPC) Approach — First, identify patient priorities, and second align care received with those priorities.
  Arms: Patient Priorities Care (PPC) Adaptation
Behavioral: Adapted PPC — First, identify patient priorities, and second align care received with those priorities.
  Arms: PPC Feasibility Testing

SUMMARY:
Most persons living with dementia (PlwD) have multiple chronic conditions (MCC). Managing MCC typically involves adhering to clinical practice guidelines for single diseases. This approach often results in burdensome care that usually does not reflect what matters most to patients. To address the challenges of caring for patients with MCC, Patient Priorities Care (PPC) was developed - a process that aligns treatment recommendations with patient priorities rather than single-disease guidelines, to improve care. Successful completion of this pragmatic pilot project will help determine how to best embedded PPC in a Healthcare system that serves a large Hispanic population. The investigators will determine if the benefits previously reported with the use of PPC hold in Hispanics with dementia.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

* Primary Objective Adapt PPC to be culturally appropriate for Hispanics with dementia and test its feasibility in an outpatient setting.
* Secondary Objectives The adapted version of PPC will improve care by identifying the healthcare priorities of Hispanics with dementia and aligning these priorities with the care participants receive.

BACKGROUND AND RATIONALE

* Background on Condition, Disease, or Other Primary Study Focus Most older adults with dementia have multiple chronic conditions (MCC), experience difficulty managing their MCC, and have poorer outcomes. Managing MCC typically involves adhering to single-disease clinical practice guidelines (CPG). This approach often results in burdensome care with outcomes that may not reflect what matters most to patients. To address the challenges for caring for patients with MCC, Patient Priorities Care (PPC) was developed - an approach that aligns disease management with patient priorities rather than CPG, to improve care. PPC is feasible and effective. Patients report less burdensome treatment and have fewer medications and referrals after going through PPC. PPC also helps clinicians recommend home and community services that are aligned with patient priorities. Focusing on patient priorities rather than CPG is a patient-centered approach that integrates well in routine clinic encounters.
* Study Rationale Physical, emotional, and cognitive impairments related to dementia interfere with disease self-management. Persons living with dementia (PlwD) therefore rely on caregivers for care and decision-making. Caregivers may add complexity to the patient-clinician interaction but are essential for translating 'what matters most' for PlwD into healthcare decisions. Patient and caregiver involvement should include identifying outcome goals and care preferences (health priorities) as well as aligning care to meet those priorities. It is therefore important to integrate caregivers into the healthcare process to achieve high-quality, family-centered care.

PlwD from minority groups experience more difficulties and poorer outcomes compared to their Non-Hispanic White (NHW) counterparts. Hispanics are the fastest-growing underrepresented population in the USA and have 1.5 times higher risk of dementia compared to NHW. Hispanics rely heavily on their families and there is a cultural expectation of families to provide care to members in need. Recent data report older Hispanics prefer care at home rather than professional care. These cultural differences and language barriers play key roles in shaping healthcare priorities and how priorities impact outcomes among Hispanics.

STUDY DESIGN For the adaptation 5 Hispanic patients will be included and for the feasibility test 20 Hispanic patients will be included.

The process will be as follows:

1. Eligible Hispanic patients will be identified through the patient roster of the Geriatrics Outpatient Clinic at UTMB.
2. Primary care providers will be asked to select patients that would not be good candidates for the study.
3. A research team member will contact the eligible patients and invite them to schedule the priority setting an appointment. For those that agree she will obtain assent and/or consent and schedule the session.
4. On the day of the session, the facilitator will use the PPC materials and identify the patient priorities, and document them in the electronic health record (Step 1). The visit will be audio recorded.
5. A research team member will schedule an appointment with the patient's primary care provider (PCP) within 2 weeks to conduct the alignment portion of the PPC approach (Step two).
6. The primary care provider will discuss the patient priorities and the provider will align care to meet those priorities and document changes in care based on the discussion on the electronic health record.
7. A research member will call the patient and assess their satisfaction with the PPC approach 2 weeks after the visit with the primary care provider.
8. A research member will contact the primary care provider and assess their satisfaction with the PPC approach.
9. The PI, Co-PI, and advisory team will review all the information and make adjustments to the protocol for the feasibility phase.
10. Activities 1-8 will be repeated with 20 Hispanic patients to test the feasibility of the adapted PPC approach for Hispanics. Given the presence of cognitive impairment, consent from a family caregiver will be obtained.

ELIGIBILITY:
Inclusion Criteria:

A) For adaptation (n=5)

* Patient's primary care provider is located in the UTMB Geriatrics Outpatient Clinic in Galveston.
* Patient identifies as Hispanic.
* Patient speaks English or Spanish.
* Patient has multiple chronic conditions listed as diagnoses in their electronic health record (3 or more chronic conditions).
* Consent to participate in all parts of the study.
* Primary care provider agrees with participation. B) For feasibility testing (n=20)
* Patient's primary care provider is located in the UTMB Geriatrics Outpatient Clinic in Galveston.
* Patient identifies as Hispanic.
* Patient speaks English or Spanish.
* Patient has multiple chronic conditions listed as diagnoses in their electronic health record (3 or more chronic conditions).
* Patient has diagnosis of dementia.
* Have a caregiver willing to participate in the study.
* Patient consent if he/she has capacity as deemed by their primary care provider or assent if he/she doesn't have capacity.
* Caregiver consent.

Exclusion Criteria:

A) For adaptation (n=5)

* Patient's primary care provider located at UTMB but not in the Geriatrics Outpatient Clinic.
* Non-Hispanic patients.
* Speaks language other than English or Spanish.
* Patient does not have multiple chronic conditions.
* Deemed ineligible by primary care provider.
* Patient has diagnosis of dementia. B) For feasibility testing (n=20)
* Patient's primary care provider located at UTMB but not in the Geriatrics Outpatient Clinic.
* Non-Hispanic patients.
* Speaks language other than English or Spanish.
* Patient does not have multiple chronic conditions.
* Patient doesn't have diagnosis of dementia.
* Patient deemed ineligible by primary care provider.
* Patient doesn't provide consent or assent based on capacity.
* Caregiver doesn't provide consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aanand D Naik, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Medical Branch in Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of participants and their caregivers will be made available to other researchers once results have been released to clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once results have been submitted to clinicaltrials.gov the listed materials will be available to share with other researchers.
Access Criteria: Data will be shared with researchers upon request to the Pi or Co-PI of the study.

REFERENCES:
- [Background] Tinetti ME, Costello DM, Naik AD, Davenport C, Hernandez-Bigos K, Van Liew JR, Esterson J, Kiwak E, Dindo L. Outcome Goals and Health Care Preferences of Older Adults With Multiple Chronic Conditions. JAMA Netw Open. 2021 Mar 1;4(3):e211271. doi: 10.1001/jamanetworkopen.2021.1271. PMID 33760091
- [Background] Freytag J, Dindo L, Catic A, Johnson AL, Bush Amspoker A, Gravier A, Dawson DB, Tinetti ME, Naik AD. Feasibility of Clinicians Aligning Health Care with Patient Priorities in Geriatrics Ambulatory Care. J Am Geriatr Soc. 2020 Sep;68(9):2112-2116. doi: 10.1111/jgs.16662. Epub 2020 Jul 20. PMID 32687218
- [Background] Tinetti ME, Naik AD, Dindo L, Costello DM, Esterson J, Geda M, Rosen J, Hernandez-Bigos K, Smith CD, Ouellet GM, Kang G, Lee Y, Blaum C. Association of Patient Priorities-Aligned Decision-Making With Patient Outcomes and Ambulatory Health Care Burden Among Older Adults With Multiple Chronic Conditions: A Nonrandomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1688-1697. doi: 10.1001/jamainternmed.2019.4235. PMID 31589281
- [Background] Blaum CS, Rosen J, Naik AD, Smith CD, Dindo L, Vo L, Hernandez-Bigos K, Esterson J, Geda M, Ferris R, Costello D, Acampora D, Meehan T, Tinetti ME. Feasibility of Implementing Patient Priorities Care for Older Adults with Multiple Chronic Conditions. J Am Geriatr Soc. 2018 Oct;66(10):2009-2016. doi: 10.1111/jgs.15465. Epub 2018 Oct 3. PMID 30281777
- [Background] Naik AD, Dindo LN, Van Liew JR, Hundt NE, Vo L, Hernandez-Bigos K, Esterson J, Geda M, Rosen J, Blaum CS, Tinetti ME. Development of a Clinically Feasible Process for Identifying Individual Health Priorities. J Am Geriatr Soc. 2018 Oct;66(10):1872-1879. doi: 10.1111/jgs.15437. Epub 2018 Oct 3. PMID 30281794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on Hispanic ethnicity from a UTMB Galveston outpatient clinic, participants without cognitive impairment, and with cognitive impairment. The first participant was enrolled on May 31st, 2022 and the last participant was enrolled in January 2024.
Pre-assignment Details: The number of participants started/completed represents the number of individual participants.
Groups:
- Patient Priorities Care (PPC) Adaptation: Participants are Hispanic patients with multiple chronic conditions (MCC) and no dementia. Participants went through two parts of the Patient Priorities Care (PPC) approach: 1) Priority Setting; and 2) Care Alignment
- PPC Feasibility Testing: Participants are Hispanics participants diagnosed mild cognitive impairment or dementia and multiple chronic conditions (MCC) were recruited. They went through two parts of the Patient Priorities Care (PPC) approach: 1) Priority Setting; and 2) Care Alignment
Period: Overall Study
Arm/Group | Patient Priorities Care (PPC) Adaptation | PPC Feasibility Testing
Started | 5 | 16
Completed | 4 | 14
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants from the adaptation phase were different from those in the feasibility phase. Baseline Characteristics were not collected for caregivers.
Groups:
- PPC Adaptation: Five participants with multiple chronic conditions
- PPC Feasibility: Sixteen with multiple chronic conditions and cognitive impairment
- Total: Total of all reporting groups
Arm/Group | PPC Adaptation | PPC Feasibility | Total
Number analyzed (Participants) | 5 | 16 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 16 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 11 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 16 | 21
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 16 | 21
Cognitive impairment [Count of Participants; unit: Participants] — The Montreal Cognitive Assessment (MoCA) - is a validated tool for cognitive screening. We used the version validated for assessments on the phone and we used the validated Spanish Version. If a MoCA score was below 8, the participants was deemed unable to consent for themselves and the caregiver was asked to consent for them, while the participants provided verbal assent.
  Participants | 0 | 16 | 16
Multiple Chronic Conditions [Count of Participants; unit: Participants] — Participants with more than 2 chronic conditions identified in their medical record
  Participants | 5 | 16 | 21

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Perceived Value of Patient Priorities Care (PPC) Approach
Description: Participants were asked to grade how valuable they thought the PPC approach was. We report the percentage of participants who responded "valuable" or "very valuable" on a scale from 1 to 5 with 1 representing "not valuable" and 5 representing "very valuable".
Time Frame: On average one month after baseline
Population: One participant from the Adaptation arm was lost to follow-up after the initial visit. In the Feasibility testing group one participant withdrew after consenting and before the first visit, and one participant was lost to follow-up after completing the intervention. Only patients are included in the analysis, caregivers are not active participants in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Patient Priorities Care (PPC) Adaptation | PPC Feasibility Testing
Number analyzed (Participants) | 4 | 14
percentage of participants | 75 | 85.7

2. Secondary Outcome: Number of Participants With Documented Changes in the Electronic Health Record That Indicate Care Alignment Was Done
Description: Dichotomous variable (yes vs no). Review of medical records to identify changes in care based on priorities identified by participants as a result of the Patient Priorities Care (PPC) approach. All medical charts were reviewed for language indicating that the primary care providers used the patient priorities to align the care provided to the patient. The default sentence provided to the providers was "Based on the patient's specific priorities, including outcome goals and care preferences, we decided to..." If information resembling this wording was found, then Care alignment was marked as positive. Otherwise, it was marked as negative.
Time Frame: Approximately one month after baseline
Population: One participant was lost to follow-up after baseline and did not complete the study in the Adaptation group. In the feasibility group one participants withdrew before the PPC approach could be completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Priorities Care (PPC) Adaptation | PPC Feasibility Testing
Number analyzed (Participants) | 5 | 16
Participants | 4 | 15

ADVERSE EVENTS:
Time Frame: 18 months
Description: 1 participant from the adaptation and feasibility group did not complete the intervention. Hence, we did not assess adverse events in them.
Arm/Group | Patient Priorities Care (PPC) Adaptation | PPC Feasibility Testing
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 0/4 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT05303194/Prot_SAP_000.pdf